CLINICAL TRIAL: NCT03256708
Title: Double-blind Randomised Placebo-controlled Study of Prolardii Gastro-resistant (GR) Caps in the Prevention and Treatment of Antibiotic-associated Diarrhoea.
Brief Title: Prevention of Antibiotic-Associated Diarrhoea With Prolardii
Acronym: PAADI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Therabel Pharma SA/NV (Industry)
Collaborators: ECSOR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: THE-2017-001
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: antibiotic-associated diarrhea; probiotic; prebiotic; placebo; synbiotic

STUDY DESIGN:
Intervention Model Description: Double-blind parallel placebo-controlled randomized study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolardii (Experimental): Prolardii GR Caps includes 4 strains of living lyophilized lactic bacteria (Lactobacillus rhamnosus GG, Bifidobacterium lactis B94, Lactobacillus casei 5773 and Lactobacillus acidophilus LA3), a yeast (Saccharomyces boulardii), a fructo-oligosaccharide (Actilight) and a dry extract of Inula helenium.
  Interventions: Dietary Supplement: Prolardii
- Placebo (Placebo Comparator): Inactive ingredients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prolardii — Prolardii: 2 capsules per day for 12 to 15 days
  Arms: Prolardii
Dietary Supplement: Placebo — Inactive ingredients
  Arms: Placebo

SUMMARY:
Prolardii contains intestinal bacteria, a yeast, a fructo-oligosaccharide and a plant extract that can contribute to the intestinal comfort. This product could prevent the diarrhea which sometimes occurs when the patient has to take antibiotics.

A total of 220 patients being prescribed antibiotics by general practitioners will be included in the study and randomized into a Prolardii arm and a placebo arm.

The primary endpoint will be the overall frequency of diarrhea in the two treatment groups. Acute diarrhea will be defined as the presence of three or more abnormally loose or watery stools per day.

DETAILED DESCRIPTION:
Prolardii is a synbiotic (prebiotic and probiotic) formulation including 4 strains of living lyophilized lactic bacteria (Lactobacillus rhamnosus GG, Bifidobacterium lactis B94, Lactobacillus casei 5773 and Lactobacillus acidophilus LA3), a yeast (Saccharomyces boulardii), a fructo-oligosaccharide (Actilight) and a dry extract of Inula helenium, a plant that can contribute to the intestinal comfort.

Taking into account the international literature, we made the assumption that the combination of probiotics and prebiotics into the same synbiotic product could improve the prevention of antibiotic-associated diarrhea and could also attenuate the intestinal symptoms related to the use of antibiotics. According to our knowledge this association has never been tested in a double-blind, randomised, placebo-controlled study.

The study will be double-blind, parallel-group, randomized, multicentre and placebo-controlled. A total of 220 patients being prescribed broad-spectrum antibiotics by general practitioners will be included in the study and randomized (1:1) into a Prolardii arm (2 capsules per day for 12 to 15 days) and a placebo arm (2 capsules per day for 12 to 15 days). There will be two medical visits (baseline visit and end-of-treatment visit) and one follow-up phone call (4 weeks after the end of treatment). During the treatment, the patients will filled in a diary card on a daily basis. They will record the number of bowel movements, the quality of the stools, the solicited symptoms (flatulence, bloating, abdominal pain/cramps, nausea and vomiting), their quality of life and the use of concomitant medications.

The data will be collected in an electronic case report form. The sample size calculation was based on the following assumptions: an attack rate in the placebo group situated in a range between 20% and 25%, an efficacy of Prolardii of about 60%, a randomization ratio 1:1 between the placebo and the active treatment group, a power of 80% and a Type I error value of 5%. Taking into account these assumptions a total of at least 30 diarrhoea cases should be reached all together in the two treatment groups, in order to ensure a sufficient power.

The primary endpoint will be the overall frequency of diarrhea in the two treatment groups. Acute diarrhea will be defined as the presence of three or more abnormally loose or watery stools per day.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female patient
* Patient aged 18 to 65 years-old
* Patient being prescribed broad spectrum antibiotics for a minimum period of 7 days and a maximum period of 10 days. Broad spectrum antibiotics are aminopenicillins (amoxicillin with or without clavulanic acid, ampicillin), cephalosporins (cefadroxil, cephalexin, cefazolin, cefuroxime, cefotaxime, ceftazidime, ceftriaxone and ceftaroline), fluoroquinolones (ciprofloxacin, levofloxacin, moxifloxacin, norfloxacin), tetracyclines (doxycycline, minocycline), nitrofurans (nitrofurantoin) and/or antibacterial sulfonamides (co-trimoxazol).
* Patient who the investigator believes that they can and will comply with the requirements of the protocol.

Exclusion Criteria:

* Patient treated with antibiotics within 3 months before inclusion in the study
* Pregnant or lactating woman
* Woman wishing to be pregnant
* Immunosuppressed subject
* Subject having a central venous catheter
* History of chronic diarrhoea
* History of irritable bowel syndrome
* History of Crohn's disease
* History of ulcerative colitis
* History of chronic constipation and/or chronic use of laxatives
* Patient with a clinically-active malignancy.
* Patient who participated in a clinical study in the previous three months
* History of psychological disorder, mental dysfunction, alcohol or drug abuse or any other factor which might interfere with the ability to cooperate in the study.
* Patient who is not sufficiently motivated to engage on a follow-up period of approximately 1.5 month, unable to complete the patient diary, or likely to travel or to move before the end of the study
* Intolerance to lactose
* Difficulty or inability to swallow '00' size capsules
* Allergy to one or several ingredients of Prolardii® GR Caps and in particular to yeasts.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Prevention of antibiotic-associated diarrhea | Antibiotic treatment duration (7 to 10 days) + 5 days
  Percentage of patients presenting an acute antibiotic-associated diarrhea

SECONDARY OUTCOMES:
Duration of diarrhea | Antibiotic treatment duration (7 to 10 days) + 5 days
  Number of days of diarrhea
Number of bowel movements | Antibiotic treatment duration (7 to 10 days) + 5 days
  Number of defecations
Tolerability of the study treatment | Antibiotic treatment duration (7 to 10 days) + 5 days
  Percentage of patients showing solicited symptoms (flatulence, bloating, abdominal pain/cramps, nausea and/or vomiting)
Quality of life of the patients | Antibiotic treatment duration (7 to 10 days) + 5 days
  Quality of life score
Safety of the study treatment | Antibiotic treatment duration (7 to 10 days) + 5 days
  Percentage of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Foucart, Study Director — Marketing Manager
Locations (1):
- ResearchLink, Linkebeek, Belgium

IPD SHARING:
Plan to Share IPD: No